CLINICAL TRIAL: NCT05052138
Title: Effects of Tactile Massage in Improving Older Residents' Psychological Health and Related Indicators in Long-Term Care Facilities
Brief Title: Effects of Tactile Massage in Long-Term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N202002045
Record Dates: First submitted 2021-09-02; First posted 2021-09-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-07

CONDITIONS: Loneliness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tactile massage (Experimental): Tactile massage 1 will receivetwo 15-min tactile massages (hand massage) per week for 4 weeks
  Interventions: Other: Tactile massage
- comparison group (No Intervention): The comparison group will receive regular care and activities.

INTERVENTIONS:
Other: Tactile massage — Tactile massage will receive two 15-min tactile massages(hand massage) per week for 4weeks
  Arms: Tactile massage

SUMMARY:
The older residents in the long-term care facilities frequently experience loneliness, anxiety, and depressive symptoms. Improving residents' psychological health problems is one of the important tasks for nursing staff. Individual experiences a sense of security and feels of being cared for after tactile massage (TM).The randomized controlled trial research design and convenience sampling will be employed. Through skin-to-skin contact, the oxytocin can be induced to make individual feel relaxed, reduce anxiety, and feel pleasure. The randomized controlled trial research design and convenience sampling will be employed. The eligible residents will be randomly assigned to intervention group and comparison group (usual care). The intervention group will receive two 15-min tactile massages per week for 4 weeks. The comparison group will receive regular care and activities.

DETAILED DESCRIPTION:
The older residents in the long-term care facilities frequently experience loneliness, anxiety, and depressive symptoms. The negative emotions might affect residents' quality of life and even increase their mortality. Improving residents' psychological health problems is one of the important tasks for nursing staff. Individual experiences a sense of security and feels of being cared for after tactile massage (TM). Through skin-to-skin contact, the oxytocin can be induced to make individual feel relaxed, reduce anxiety, and feel pleasure. Moreover, TM does not need any tools and can be conducted at any time and any place. It is very convenient and accessible. Therefore, the purpose of this study is going to examine the effects of tactile massage in improving older residents' mental health and physiological effect in LTCFs. The randomized controlled trial research design and convenience sampling will be employed. LTCFs will be selected and contacted by researchers. The eligible residents will be randomly assigned to intervention group and comparison group (usual care). The intervention group will receive two 15-min tactile massages per week for 4 weeks. The comparison group will receive regular care and activities. Data will be collected at baseline, after intervention using questionnaires including demographic and related information questionnaire, University of California Los Angeles (UCLA) loneliness Scale version 3, Geriatric Anxiety Inventory, Geriatric Depression Scale short form (GDS-SF).Chinese Happiness Inventory, comfort Visual Analogue Scale, Relaxed Visual Analogue Scale, and vital signs. Data analysis will be conducted by performing percentage, mean, t-test, chi-square, and generalized estimating equations (GEE) using SPSS 22.0 software. Intention-to-treat analysis will be applied in this study.

ELIGIBILITY:
Inclusion Criteria:

* have lived in long-term care facilities for over one month
* conscious clear and can clearly express him or herself.

Exclusion Criteria:

* infection disease and skin problems
* psychiatric disorders
* loss sense of both hands.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
University of California Los Angeles (UCLA)loneliness Scale version 3 | baseline, pre-intervention(T0)
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from 1 (Never) to 4 (Often). The total score ranged 20~80 points, with a higher score indicating high level of loneliness
University of California Los Angeles (UCLA)loneliness Scale version 3 | after the completion of the intervention(T1)
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from 1 (Never) to 4 (Often). The total score ranged 20~80 points, with a higher score indicating high level of loneliness
Geriatric Depression Scale short form (GDS-SF) | baseline, pre-intervention(T0)
  The Geriatric Depression Scale is a 15-item "yes/no" self-report measure of depressive symptom.The individual is asked to report whether they have experienced these symptoms over the past week. The Geriatric Depression Scale has a maximum score of 15, with higher scores representing more severe symptoms.
Geriatric Depression Scale short form (GDS-SF) | after the completion of the intervention(T1)
  The Geriatric Depression Scale is a 15-item "yes/no" self-report measure of depressive symptom.The individual is asked to report whether they have experienced these symptoms over the past week. The Geriatric Depression Scale has a maximum score of 15, with higher scores representing more severe symptoms.
Geriatric Anxiety Inventory (GAI) | baseline, pre-intervention(T0)
  The Geriatric Anxiety Inventory is a 20-item "yes/no" self-report measure of Anxiety symptom.The individual is asked to report whether they have experienced these symptoms over the past week. The Geriatric Anxiety Inventory has a maximum score of 20, with higher scores representing more severe symptoms.
Geriatric Anxiety Inventory (GAI) | after the completion of the intervention(T1)
  The Geriatric Anxiety Inventory is a 20-item "yes/no" self-report measure of Anxiety symptom.The individual is asked to report whether they have experienced these symptoms over the past week. The Geriatric Anxiety Inventory has a maximum score of 20, with higher scores representing more severe symptoms.
body temperature(BT) | baseline, pre-intervention(T0)
  body temperature use ear thermometer measure temperature，normal body temperature can range between 36.1 C and 37.2 C .
body temperature(BT) | through study completion, an average of 1 weeks(T1)
  body temperature use ear thermometer measure temperature，normal body temperature can range between 36.1 C and 37.2 C .
body temperature(BT) | through study completion,week 2 (T2)
  body temperature use ear thermometer measure temperature，normal body temperature can range between 36.1 C and 37.2 C .
body temperature(BT) | through study completion, week 3 (T3)
  body temperature use ear thermometer measure temperature，normal body temperature can range between 36.1 C and 37.2 C .
body temperature(BT) | after the completion of the intervention(T4)
  body temperature use ear thermometer measure temperature，normal body temperature can range between 36.1 C and 37.2 C .
blood pressure(BP) | baseline, pre-intervention(T0)
  Upper Arm blood pressure monitor measure, blood pressure is considered to be between 90/60 mmHg and 120/80 mmHg
blood pressure(BP) | through study completion, an average of 1 weeks(T1)
  Upper Arm blood pressure monitor measure, blood pressure is considered to be between 90/60 mmHg and 120/80 mmHg
blood pressure(BP) | through study completion,week 2 (T2)
  Upper Arm blood pressure monitor measure, blood pressure is considered to be between 90/60 mmHg and 120/80 mmHg
blood pressure(BP) | through study completion, week 3 (T3)
  Upper Arm blood pressure monitor measure, blood pressure is considered to be between 90/60 mmHg and 120/80 mmHg
blood pressure(BP) | after the completion of the intervention(T4)
  Upper Arm blood pressure monitor measure, blood pressure is considered to be between 90/60 mmHg and 120/80 mmHg
heart rate(HR) | baseline, pre-intervention(T0)
  measure heart rate, simply check pulse. To check your pulse at your wrist, two fingers between the bone and the tendon over your radial artery . ranges from 60 to 100 beats per minute.
heart rate(HR) | through study completion, an average of 1 weeks(T1)
  measure heart rate, simply check pulse. To check your pulse at your wrist, two fingers between the bone and the tendon over your radial artery . ranges from 60 to 100 beats per minute.
heart rate(HR) | through study completion,week 2 (T2)
  measure heart rate, simply check pulse. To check your pulse at your wrist, two fingers between the bone and the tendon over your radial artery . ranges from 60 to 100 beats per minute.
heart rate(HR) | through study completion, week 3 (T3)
  measure heart rate, simply check pulse. To check your pulse at your wrist, two fingers between the bone and the tendon over your radial artery . ranges from 60 to 100 beats per minute.
heart rate(HR) | after the completion of the intervention(T4)
  measure heart rate, simply check pulse. To check your pulse at your wrist, two fingers between the bone and the tendon over your radial artery . ranges from 60 to 100 beats per minute.
breathing rate(RR) | baseline, pre-intervention(T0)
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.
breathing rate(RR) | through study completion, an average of 1 weeks(T1)
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.
breathing rate(RR) | through study completion,week 2 (T2)
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.
breathing rate(RR) | through study completion, week 3 (T3)
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.
breathing rate(RR) | after the completion of the intervention(T4)
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.

SECONDARY OUTCOMES:
Chinese Happiness Inventory | baseline, pre-intervention(T0)
  A 10-item scale designed to measure one's subjective feelings of Happiness . Participants rate each item on a scale from 0 to 3. The total score ranged 0~30 points, with a higher score indicating high level of happy
Chinese Happiness Inventory | after the completion of the intervention(T1)
  A 10-item scale designed to measure one's subjective feelings of Happiness . Participants rate each item on a scale from 0 to 3. The total score ranged 0~30 points, with a higher score indicating high level of happy
comfort Visual Analogue Scale | baseline, pre-intervention(T0)
  providing a range of scores from 0-10. A higher score indicates greater comfort intensity
comfort Visual Analogue Scale | through study completion, an average of 1 weeks(T1)
  providing a range of scores from 0-10. A higher score indicates greater comfort intensity
comfort Visual Analogue Scale | through study completion, week 2 (T2)
  providing a range of scores from 0-10. A higher score indicates greater comfort intensity
comfort Visual Analogue Scale | through study completion, week 3 (T3)
  providing a range of scores from 0-10. A higher score indicates greater comfort intensity
comfort Visual Analogue Scale | after the completion of the intervention(T4)
  providing a range of scores from 0-10. A higher score indicates greater comfort intensity
Relaxed Visual Analogue Scale | baseline, pre-intervention(T0)
  providing a range of scores from 0-10. A higher score indicates greater Relaxed intensity
Relaxed Visual Analogue Scale | through study completion, an average of 1 weeks(T1)
  providing a range of scores from 0-10. A higher score indicates greater Relaxed intensity
Relaxed Visual Analogue Scale | through study completion, week 2 (T2)
  providing a range of scores from 0-10. A higher score indicates greater Relaxed intensity
Relaxed Visual Analogue Scale | through study completion, week 3 (T3)
  providing a range of scores from 0-10. A higher score indicates greater Relaxed intensity
Relaxed Visual Analogue Scale | after the completion of the intervention(T4)
  providing a range of scores from 0-10. A higher score indicates greater Relaxed intensity

CONTACTS AND LOCATIONS:
Overall Officials: Pi-Hua Huang, Principal Investigator — Taipei Medical University
Locations (2):
- Taiwan (2):
  - Suao Veterans Hospital, Tainan, Yilan
  - Tung Jen Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yucel SC, Arslan GG, Bagci H. Effects of Hand Massage and Therapeutic Touch on Comfort and Anxiety Living in a Nursing Home in Turkey: A Randomized Controlled Trial. J Relig Health. 2020 Feb;59(1):351-364. doi: 10.1007/s10943-019-00813-x. PMID 30982141
- [Background] Nakano H, Kodama T, Ueda T, Mori I, Tani T, Murata S. Effect of Hand and Foot Massage Therapy on Psychological Factors and EEG Activity in Elderly People Requiring Long-Term Care: A Randomized Cross-Over Study. Brain Sci. 2019 Mar 4;9(3):54. doi: 10.3390/brainsci9030054. PMID 30836612
- [Background] Kunikata H, Watanabe K, Miyoshi M, Tanioka T. The effects measurement of hand massage by the autonomic activity and psychological indicators. J Med Invest. 2012;59(1-2):206-12. doi: 10.2152/jmi.59.206. PMID 22450009
- [Background] McFeeters S, Pront L, Cuthbertson L, King L. Massage, a complementary therapy effectively promoting the health and well-being of older people in residential care settings: a review of the literature. Int J Older People Nurs. 2016 Dec;11(4):266-283. doi: 10.1111/opn.12115. Epub 2016 Feb 15. PMID 26875503
- [Result] Suzuki M, Tatsumi A, Otsuka T, Kikuchi K, Mizuta A, Makino K, Kimoto A, Fujiwara K, Abe T, Nakagomi T, Hayashi T, Saruhara T. Physical and psychological effects of 6-week tactile massage on elderly patients with severe dementia. Am J Alzheimers Dis Other Demen. 2010 Dec;25(8):680-6. doi: 10.1177/1533317510386215. PMID 21131675
- [Derived] Huang PH, Chien WP, Lin YC, Chung MH, Lin PC, Lin YK, Chuang YH. Effects of Tactile Massage in Improving Older Residents' Psychological Health in Long-Term Care Facilities: A Randomised Controlled Trial. Int J Older People Nurs. 2024 Sep;19(5):e12652. doi: 10.1111/opn.12652. PMID 39312625

DOCUMENTS (2):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT05052138/Prot_002.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT05052138/SAP_003.pdf